CLINICAL TRIAL: NCT02323555
Title: Optimize the Requirements and Preparations in Outpatient Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPTIMA
Record Dates: First submitted 2014-08-01; First posted 2014-12-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-08

CONDITIONS: Cancer; IV Anticancer Therapy
Keywords: Cancer; chemotherapy; Targeted therapy; Day Hospital
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paramedic telephone consultation (Experimental): Establishment of a paramedic telephone consultation to the doctor to record the "virtual" early prescription or non-injectable cancer treatment before the arrival of the patient (Feasibility Process Optima), without changing the current practice of prescribing and dispensing of these treatments on the day of the coming of the patient.
  Interventions: Other: Paramedic telephone consultation

INTERVENTIONS:
Other: Paramedic telephone consultation

SUMMARY:
A prescription of injectable anticancer therapy requires the collection of medical data (interview and physical examination) and often allied (laboratory tests). This requirement is made on the day of the arrival of the patient to not prepare these treatments incorrectly.

After receiving the prescription of treatment, it will take about 1 hour to prepare for pharmacy and more in times of high activity, to provide the day hospital pockets treatment, incompressible time when the patient waits to have his treatment.

A process has been selected (Optima) to anticipate prescribing injectable cancer treatments and their manufacturing to reduce patient waiting times on the day of his coming François BaclesseCentre day hospital.

DETAILED DESCRIPTION:
Given the investigators daily activity evaluated patients received 65-70 day hospital, assessing the feasibility of the project with an internalized platform seems most relevant to completely control the process and costs.

This project will consist of anticipation paramedic telephone consultation followed by a medical prescription validation will trigger the production of chemotherapy prematurely before the coming of the patient.

The François Baclesse Center therefore supports the idea of an early day hospital, that is to say a prescription and production pockets of chemotherapy before the arrival of the patient in the service.

This project was named PROJECT OPTIMA for "Optimize requirements and preparations chemotherapy Ambulatory Medicine" with a paramedic telephone consultation.

So this ambitious project is the first experience of a French advance routine injectable anticancer therapies, all protocols combined in a Centre for the Fight against Cancer but also in a hospital reference competent oncology and chemotherapy and whose preparation process of chemotherapy administered by injection is fully internalized and centralized.

Before starting this program routine, it is essential to validate through a research project concordance between paramedic telephone consultation structured using tools and medical consultation but also define the profiles of patients and types of chemotherapy injectable likely to benefit safely from this program.

This study will be conducted in two parts:

• Part 1: where are compared two tools:

* paramedical examination conducted by telephone two days before the arrival of the patient by a trained nurse, according to a predetermined grid, as a basis for medical decisions prescription "virtual" or non-treatment;
* medical examination performed on the day of the coming of the patient for treatment.

This component will run for three months and will evaluate the rate of discrepancies between these 2 types of prescription.

During this period, any prescription or administration of treatment will be validated at the end of the paramedical examination phones.

This component will also detect and specify protocols suitable injectable cancer treatment and develop a typology of patients for whom the anticipation process is more efficient and more secure.

Indeed, the investigators can think that the anticipation process will not be effective for all patients.

For example, a patient with a brain tumor will often diminished cognitive abilities including its memory abilities. Responses to the telephone interview conducted by the nurse may be incomplete or even false due to its memory disorders.

At the same time, waiting times and patient satisfaction will be evaluated and used as a reference for the second part of the study whose objective is to evaluate the benefits of this early prescription used routinely.

• 2nd part: It is an assessment process routinely used after defining the profile of patients and types of treatment protocols, including the phone call from the nurse, the early prescription of chemotherapy, early production and day, medical consultation control before administration.

In this step will be compared to expectations time, patient satisfaction and treatment wrongly prepared before and after the launch of Optima.

Prerequisites:

* All nurses to conduct telephone interviews will be trained on two days conducted by EFEC (European School of Oncology Training) whose purpose is to explain the issues of the telephone interview for resulting prescription chemotherapy for the patient.
* Nurses phone platform dedicated to the call of patients will experience in service, allowing them to develop acuity to identify clues that signpost to important pieces of information for the management of patients.

Feasibility:

This study will be conducted in two stages for a period of three months each, which should allow in the investigators activity to include 450 patients by step, based on 3 patient came through, about 1350 came by step ..

The homepage of the day hospital service capacity is 40 places for activity 65-70 patients per day. Approximately 300 patients are admitted each week with about 42 new patients each week.

The investigators welcome all specialties outside of Hematology (digestive oncology, ENT and Pneumology, urogynecologic, breast screening, brain tumors and sarcomas).

ELIGIBILITY:
Inclusion Criteria:

* Patient (e) old (e) 18 or more;
* Patient (e) reached (e) from cancer and candidate (s) to treatment with injectable anticancer preparations in day hospital
* solid cancerous disease for which chemotherapy is given intravenously;
* Patient (e) able to communicate with the investigator or his representative;
* Patient (e) Affiliate (e) a social security scheme;
* Mastery of the French language;
* Consent and signed.

Exclusion Criteria:

* Exclusive orallyanticancer treatment ;
* Primary brain tumors;
* Patient (e) dysphonic or having difficulty communicating orally;
* Patient (e) receiving intravenous chemotherapy as part of a research protocol;
* Patient (e) to receive chemotherapy whose stability is less than 24:00 (Temsirolimus)
* Pathologies hematologic malignancies
* Inability to undergo medical monitoring test for geographical, social or psychological reasons.
* Patient (e) under guardianship or unable to give informed consent;
* Patient (s) whose cognitive functions do not allow a telephone interview.
* Any medical or psychological condition associated that could compromise the patient's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patient profile for Optima | up to 21 weeks
  Rate of discordance for each chemotherapy protocol between the Optima process and the current process.
  Define which protocols for injectable cancer treatment (chemotherapy and / or targeted therapy) and for which patient profiles, the Optima process can be used routinely.

SECONDARY OUTCOMES:
Satisfaction | up to 21 weeks
  Patient satisfaction will be collected through the questionnaire OUTPATSAT 35

CONTACTS AND LOCATIONS:
Overall Officials: Audrey FAVEYRIAL, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François Baclese, Caen, France